CLINICAL TRIAL: NCT02051270
Title: Mild Cognitive Impairment and Balance in Elderly
Brief Title: Cognitive Impairment and Balance in Elderly
Status: Completed | Type: Observational
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, assistant professor, Universidad de Granada
Other Study IDs: DF0050UG
Record Dates: First submitted 2014-01-27; First posted 2014-01-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Mild Cognitive Impairment
Keywords: Elderly; Nursing homes; Mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Elders: Older people living in nursing homes will undergo a descriptive study.
  Interventions: Other: Descriptive study

INTERVENTIONS:
Other: Descriptive study — More than 65 years old elders

SUMMARY:
One important issue in older adults with cognitive problems is the higher risk of fall due to decreased motor function and balance. The objective of this study is to evaluate the repercussions of mild cognitive impairment in balance in elderly.

DETAILED DESCRIPTION:
Mild cognitive impairment is described as a transitional stage between normal ageing and dementia, and reflects the clinical situation where a person has memory complaints and objective evidence of cognitive impairment but no evidence of dementia. Mild cognitive is important in older people and it is also important to evaluate its repercussion in balance.

ELIGIBILITY:
Inclusion Criteria:

* Nursing home residents.

Exclusion Criteria:

* Surgery on lower limbs.
* Traumatic damage on lower limbs.
* Severe cognitive impairment in order not to complete the assessment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elders
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Dynamic balance | baseline
  Dynamic balance is going to be measured using the Mini-Best test. This is a 14-item test that focuses on dynamic balance, specifically anticipatory transitions, postural responses, sensory orientation, and dynamic gait

SECONDARY OUTCOMES:
Cognitive impairment | baseline
  The cognitive impairment will be measured using the Montreal Cognitive Assessment and the Mini-Mental State Examination. The Montreal Cognitive Assessment is a test designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The Mini Mental State Examination is a 10-minute bedside measure of impaired thinking in undeveloped, uneducated, diseased, or very old populations.
Attention | baseline
  Attention is going to be measured with the Stroop test.
Cognitive flexibility | baseline
  The cognitive flexibility of patients is measured using the Trial Making Test. This test explores visual-conceptual and visual-motor tracking, and it is a frequently used neuropsychological test.

CONTACTS AND LOCATIONS:
Overall Officials: Marie Carmen Valenza, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Faculty of health Sciences. University of Granada, Granada, Spain, Spain

REFERENCES:
- [Background] Diaz-Pelegrina A, Cabrera-Martos I, Lopez-Torres I, Rodriguez-Torres J, Valenza MC. [Effects of cognitive state on balance disturbances and gait disorders in institutionalised elderly]. Rev Esp Geriatr Gerontol. 2016 Mar-Apr;51(2):88-91. doi: 10.1016/j.regg.2015.07.014. Epub 2015 Nov 2. Spanish. PMID 26541310